CLINICAL TRIAL: NCT02059148
Title: Effect of Food on the Pharmacokinetics of LY2835219 in Healthy Subjects
Brief Title: A Study of LY2835219 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15175; I3Y-MC-JPBG (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2835219 Standard (Experimental): Single oral dose of LY2835219 given with a standard meal in one of three study periods.
  Interventions: Drug: LY2835219
- LY2835219 Fasted (Experimental): Single oral dose of LY2835219 given with no food in one of three periods.
  Interventions: Drug: LY2835219
- LY2835219 High-Fat (Experimental): Single oral dose of LY2835219 given with a high fat meal in one of three periods.
  Interventions: Drug: LY2835219

INTERVENTIONS:
Drug: LY2835219 — Administered orally.
  Other Names: abemaciclib

SUMMARY:
Participants in this study will receive 3 single oral doses of LY2835219 at least 14 days apart. One dose will be given with a standard meal, one dose with a high-fat meal and one dose without food. The study will evaluate the effects of the standard and high-fat meals on how much drug gets into the bloodstream. Side effects will be documented. This study is approximately 43 days, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy sterile males or surgically sterile or postmenopausal females
* Have a body mass index (BMI) of 18 to 32 kilogram per meter square (kg/m^2), inclusive, at screening
* Are able to eat a high-fat, high-calorie meal

Exclusion Criteria:

* Participated in a clinical trial involving investigational product within 30 days
* Abnormal blood pressure
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have donated blood of more than 500 milliliter (mL) within the last month
* Show evidence of human immunodeficiency virus, hepatitis B or hepatitis C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Single Oral Dose of 200 mg LY2835219 on 3 Occasions: Standard Meal, Fasted State, High-Fat Meal. Dosing occasions were separated by at least 14 days.
- Sequence 2: Single Oral Dose of 200 mg LY2835219 on 3 Occasions: Standard Meal, High-Fat Meal, Fasted State. Dosing occasions were separated by at least 14 days.
- Sequence 3: Single Oral Dose of 200 mg LY2835219 on 3 Occasions: Fasted State, High-Fat Meal, Standard Meal. Dosing occasions were separated by at least 14 days.
- Sequence 4: Single oral dose of 200 mg LY2835219 on 3 Occasions: Fasted State, Standard Meal, High-Fat Meal. Dosing occasions were separated by at least 14 days.
- Sequence 5: Single oral dose of 200 mg LY2835219 on 3 Occasions: High-Fat Meal, Fasted State, Standard Meal. Dosing occasions were separated by at least 14 days.
- Sequence 6: Single Oral Dose of 200 mg LY2835219 on 3 Occasions: High-Fat Meal, Standard Meal, Fasted State. Dosing occasions were separated by at least 14 days.
Period: Treatment 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 4 | 4 | 4 | 3
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 4 | 4 | 4 | 3
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Single Oral Dose of 200 mg LY2835219 on 3 Occasions: Standard Meal, Fasted State, High-Fat Meal.
Groups:
- All Study Participants: Single Oral Dose of 200 mg LY2835219 on 3 Occasions: Standard Meal, Fasted State, High-Fat Meal. Dosing occasions were separated by at least 14 days.
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2835219 Fasted vs. High-Fat Arms
Time Frame: Predose, 0.5,1,2,3,4,6,8,10,12,24,48,72,96,120,144,168,192 hours post-LY2835219 dose in each period
Population: All randomized participants receiving at least one dose of the investigational product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | LY2835219 Fasted | LY2835219 High-Fat
Number analyzed (Participants) | 23 | 24
nanogram/milliliter (ng/mL) | 111 (61) | 137 (52)
Statistical Analysis 1: Comparison: LY2835219 Fasted vs LY2835219 High-Fat; Test type: Superiority or Other; Ratio of Geometric LSMeans = 1.24, 90% CI 2-sided [1.11 to 1.38]

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve (0-t Last) [AUC(0-t Last)] of LY2835219 Fasted vs. High-Fat Arms
Time Frame: Predose, 0.5,1,2,3,4,6,8,10,12,24,48,72,96,120,144,168,192 hours post-LY2835219 dose in each period
Population: All randomized participants receiving at least one dose of the investigational product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/mL (ng*h/mL)
Arm/Group | LY2835219 Fasted | LY2835219 High-Fat
Number analyzed (Participants) | 23 | 24
nanogram*hour/mL (ng*h/mL) | 4160 (65) | 4790 (57)
Statistical Analysis 1: Comparison: LY2835219 Fasted vs LY2835219 High-Fat; Test type: Superiority or Other; Ratio of Geometric LSMeans = 1.14, 90% CI 2-sided [1.05 to 1.23]

3. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Concentration (Tmax) of LY2835219 Fasted vs. High-Fat Arms
Time Frame: Predose, 0.5,1,2,3,4,6,8,10,12,24,48,72,96,120,144,168,192 hours post-LY2835219 dose in each period
Population: All randomized participants receiving at least one dose of the investigational product.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | LY2835219 Fasted | LY2835219 High-Fat
Number analyzed (Participants) | 23 | 24
hour (h) | 8.00 [6.00 to 12.00] | 10.00 [6.00 to 24.00]
Statistical Analysis 1: Comparison: LY2835219 Fasted vs LY2835219 High-Fat; Test type: Superiority or Other; p = 0.0006, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.95, 90% CI 2-sided [1.00 to 2.00]

4. Secondary Outcome: Pharmacokinetics: Cmax of LY2835219 in Standard Meal Arm
Time Frame: Predose, 0.5,1,2,3,4,6,8,10,12,24,48,72,96,120,144,168,192 hours post-LY2835219 dose in each period
Population: All randomized participants receiving at least one dose of the investigational product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- LY2835219 Standard: Single oral dose of LY2835219 given with a standard meal in one of three study periods.
  LY2835219 administered orally.
Arm/Group | LY2835219 Standard
Number analyzed (Participants) | 22
ng/mL | 141 (55)

5. Secondary Outcome: Pharmacokinetics: AUC(0-tlast) of LY2835219 in Standard Meal Arm
Time Frame: Predose, 0.5,1,2,3,4,6,8,10,12,24,48,72,96,120,144,168,192 hours post-LY2835219 dose in each period
Population: All randomized participants receiving at least one dose of the investigational product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | LY2835219 Standard
Number analyzed (Participants) | 22
ng*h/mL | 4610 (65)

6. Secondary Outcome: Pharmacokinetics: Tmax of LY2835219 in Standard Meal Arm
Time Frame: Predose, 0.5,1,2,3,4,6,8,10,12,24,48,72,96,120,144,168,192 hours post-LY2835219 dose in each period
Population: All randomized participants receiving at least one dose of the investigational product.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | LY2835219 Standard
Number analyzed (Participants) | 22
hour (h) | 8.00 [6.00 to 10.00]

7. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC 0-t Last) of LSN3106726 (M20)
Description: Area under the concentration versus time curve from time zero to time t, where t is the last time point with a measurable concentration of LSN3106726 (M20), an active metabolite of LY2835219.
Time Frame: Predose, 0.5,1,2,3,4,6,8,10,12,24,48,72,96,120,144,168,192 hours post-LY2835219 dose in each period
Population: All randomized participants receiving at least one dose of the investigational product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | LY2835219 Standard | LY2835219 Fasted | LY2835219 High-Fat
Number analyzed (Participants) | 22 | 23 | 24
ng*h/mL | 3590 (35) | 3320 (40) | 3510 (35)

ADVERSE EVENTS:
Arm/Group | LY2835219 Standard | LY2835219 Fasted | LY2835219 High-Fat
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 4/23 | 6/23 | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2835219 Standard (N=23) | LY2835219 Fasted (N=23) | LY2835219 High-Fat (N=24)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days